CLINICAL TRIAL: NCT04655950
Title: SPONDIMMO : Multicentered Descriptive Prospective Study of Immobilization and Neurological Complication in Patients With Vertebral Osteomyelitis.
Brief Title: Immobilization and Neurological Complications in Patients With Vertebral Osteomyelitis.
Acronym: SPONDIMMO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0214
Record Dates: First submitted 2020-02-04; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Vertebral Osteomyelitis; Spondylodiscitis
Keywords: Vertebral Osteomyelitis; Spine Immobilization; Neurological complications
MeSH Terms: conditions — Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: protocols and practices for the immobilization of vertebral osteomyelitis in different French hospitals and bone and joint infections Centers — Evaluation of the frequency of neurological complications in a large prospective cohort, and to identify clinical and imaging risk factors for neurological complications.
  We search for association between type and duration of spine immobilization and neurological status at the end of follow-up

SUMMARY:
Vertebral osteomyelitis is an infection of the intervertebral disk and adjacent vertebral plates with a non-negligible risk of neurological complications and handicap. If there are clear recommendations dealing with antibiotic therapy and surgery indications for this pathogen, the question of the immobilization will be remaining debate. The aim of the study was to describe protocols and practices for the immobilization of vertebral osteomyelitis in different French hospitals and bone and joint infections Centers. The secondary objectives were to evaluate the frequency of neurological complications in a large prospective cohort, and to identify clinical and imaging risk factors for neurological complications.

The investigators also aim to search for association between type and duration of spine immobilization and neurological status at the end of follow-up.

DETAILED DESCRIPTION:
Study design is descriptive, prospective, multicentric, and the investigators have a single database centralized in Nantes University Hospital. Patient's data will be conserved and trapped anonymously and patients all give oral consent. Information letter is given to each patient.

Typical study calendar :

Baseline :

* Patient information (letter and oral consent)
* Clinical data and comorbidities collection
* Neurological examination
* Spine X-ray
* MRI or CT-scan imaging to confirm diagnosis

During Hospitalization

* Date collection : spine immobilization modalities (type, duration, changes…), duration of bed rest
* Other treatments (antibiotic therapy : molecules and duration)
* Daily neurological examination

  3 months follow-up visit : (if usually done by physician)
* Clinical and neurological examination
* Spine immobilization assessment
* Spine X-ray
* Oswestry questionary

  6 months follow-up visit : finale visit (if usually done by physician)
* Clinical and neurological examination
* Spine immobilization assessment
* Spine X-ray
* Oswestry questionary

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, male and female
* Hospitalized of a vertebral osteomyelitis in one of the Centers
* Meeting the criteria for the definition of vertebral Osteomyelitis (typical imaging findings)
* Microbiological proof of infection (blood culture or discovertebral biopsy) or high suspicion of infection (Compatible histology, good response to antibiotics and no differential diagnosis).

Exclusion Criteria:- Spine device infection

* Recent spinal surgery less than 1month
* Children under 18 years old
* Under guardianship
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Baseline :
  * Patient information (letter and oral consent)
  * Clinical data and comorbidities collection
  * Neurological examination
  * Spine X-ray
  * MRI or CT-scan imaging to confirm diagnosis
  During Hospitalization
  * Date collection : spine immobilization modalities (type, duration, changes…), duration of bed rest
  * Other treatments (antibiotic therapy : molecules and duration)
  * Daily neurological examination
    3 months follow-up visit : (if usually done by physician)
  * Clinical and neurological examination
  * Spine immobilization assessment
  * Spine X-ray
  * Oswestry questionnary
    6 months follow-up visit : finale visit (if usually done by physician)
  * Clinical and neurological examination
  * Spine immobilization assessment
  * Spine X-ray
  * Oswestry questionnary
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Qualitative description of main types of spine immobilization | inclusion
  Type of bracing : smooth or rigid bracing, highness of bracing (cervical, thoracic, lumbar spine or both and level of the highest and lowest vertebrae included).

SECONDARY OUTCOMES:
Frequency of neurological complications | inclusion, month 3 and month 6
  Percentage of neurological complication at baseline, 3 and 6 months follow-up)
  * Percentage of major neurological signs (sphincter dysfunction and/or motor deficit and ASIA score) at baseline, 3 and 6 months follow-up
  * Percentage of minor neurological signs (radicular pain, reflex abolition, hypoesthesia) at baseline, 3 and 6 months follow-up
MRI signs at baseline | inclusion, month 3 and month 6
  Number of vertebrae involved, destruction of posterior arch, destruction of vertebrae, kyphosis, epidural phlegmon, spinal cord hypersignal, dural sac compression, anterior effacement of subarachnoidal space
  Oswestry functional score at 3 and 6 months follow-up. Association between type and duration of spine immobilization and neurological complication
Oswestry functional score at 3 and 6 months follow-up | inclusion, month 3 and month 6
  Association between type and duration of spine immobilization and neurological complication
Duration of Spine immobilization | month 6
  Evaluation of the duration of immobilization of the spine

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Le Goff, PH, Principal Investigator — Nantes University Hospital
Locations (9):
- France (9):
  - Angers University Hospital, Angers
  - Clermont ferrand University Hospital, Clermont-Ferrand
  - La Roche Sur Yon Hospital, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - Paris University Hospital, Paris
  - Quimper Hospital, Quimper
  - Rennes University Hospital, Rennes
  - Saint-Nazaire Hospital, Saint-Nazaire
  - Tours University Hospital, Tours